CLINICAL TRIAL: NCT04210713
Title: Characterization of Neuroimmune Dysfunction in Alcohol Use Disorder
Brief Title: Neuroimmune Dysfunction in Alcohol Use Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Daniel Roche, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00080891; 5K01AA026005-03 (NIH)
Record Dates: First submitted 2019-12-17; First posted 2019-12-26 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Alcohol Drinking; Alcohol-Related Disorders; Disease; Inflammation; Alcoholism; Cognitive Dysfunction; Pathologic Processes; Drinking Behavior; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorder; Cognition Disorder; Neurocognitive Disorders; Minocycline; Anti-Bacterial Agents; Anti-Infective Agents
Keywords: Minocycline
MeSH Terms: conditions — Alcohol Drinking; Alcohol-Related Disorders; Disease; Inflammation; Alcoholism; Cognitive Dysfunction; Pathologic Processes; Drinking Behavior; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorders; Cognition Disorders; Neurocognitive Disorders; cyclopia sequence | interventions — Minocycline; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- AUD-Minocycline (Active Comparator): Participants diagnosed with alcohol use disorder will be randomly assigned to take minocycline for 4 weeks. The randomization is double-blinded and will alternate between minocycline and placebo.
  Interventions: Drug: Minocycline
- AUD-Placebo (Placebo Comparator): Participants diagnosed with alcohol use disorder will be randomly assigned to take placebo for 4 weeks. The randomization is double-blinded and will alternate between minocycline and placebo.
  Interventions: Drug: Sugar pill
- Healthy Control-Minocycline (Active Comparator): Healthy control participants will be randomly assigned to take minocycline for 4 weeks. The randomization is double-blinded and will alternate between minocycline and placebo.
  Interventions: Drug: Minocycline
- Healthy Control-Placebo (Placebo Comparator): Healthy control participants will be randomly assigned to take placebo for 4 weeks. The randomization is double-blinded and will alternate between minocycline and placebo.
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Minocycline — 200 mg/day
  Arms: AUD-Minocycline; Healthy Control-Minocycline
Drug: Sugar pill — Matched placebo
  Other Names: Placebo
  Arms: AUD-Placebo; Healthy Control-Placebo

SUMMARY:
The objective of this proposal is to advance medication development for alcohol use disorder by examining the efficacy and mechanisms of action of minocycline, a neuroimmune modulator, as a potential treatment. This study has important clinical implications, as the available treatments for alcohol use disorder are only modestly effective and testing novel medications is a high research priority.

DETAILED DESCRIPTION:
The research objective of this project is to characterize the role of the neuroimmune system in alcohol use disorder (AUD). The proposed study employs a randomized, double-blind, and placebo-controlled design to examine how neuroinflammation, as measured via neuroimaging [e.g., magnetic resonance imaging (MRI)], relates to alcohol craving, neurocognitive impairment (e.g., memory, attention, etc.), and alcohol use in non-treatment seeking individuals with AUD. The study will also determine whether minocycline (MINO), an FDA-approved antibiotic medication, affects any of the above listed measures. In the proposed study, healthy controls (n = 36) and non-treatment seeking individuals with a current Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 AUD diagnosis (n = 36) will be randomized to receive either 200 mg of minocycline per day or placebo for approximately 28 days and complete two laboratory sessions. The first laboratory session will be performed immediately before commencing the medication regimen (day 0) and the second will be completed after taking the medication daily for approximately 28 days. Within each laboratory session, participants will complete a cue reactivity paradigm, neurocognitive performance tasks, and a magnetic resonance imaging (MRI) session. Additionally, blood samples will be drawn on days 0, 7, 14, 21, and 28 of treatment to measure circulating levels of proinflammatory molecules in order to identify the specific immune signaling pathways underlying neuroinflammation in AUD. Clinical labs (e.g., blood chemistry, liver function tests) and adverse events (AEs) will also be assessed at these five visits.

ELIGIBILITY:
AUD Group Inclusion Criteria:

* Meet DSM-5 diagnostic criteria for an AUD
* In the 30-day period before enrollment, consume ≥ 14 and ≥ 7 standard drinks per week for men and women, respectively, AND
* In the 30-day period before enrollment, engage in heavy drinking (5 or more drinks for men, 4 or more drinks for women) and ≥ 5 times per month

AUD Group Exclusion Criteria:

* Currently in treatment for AUD, a history of treatment within the 30 days before enrollment, or currently seeking immediate treatment
* Current (last 12 months) DSM-5 diagnosis of substance use disorder for any psychoactive substances other than alcohol and nicotine
* Currently prescribed a psychotropic medication for the treatment of schizophrenia spectrum and other psychotic disorders, bipolar and related disorders, depressive disorders, anxiety disorders, and mood disorders.
* Lifetime DSM-5 diagnosis of schizophrenia spectrum and other psychotic disorders and bipolar and related disorders
* Positive urine toxicology screen for the following substances: cocaine, opiates, amphetamines, methamphetamine, phencyclidine, barbiturates, benzodiazepine, methadone, and tricyclic antidepressants.
* Self-reported daily use of cannabidiol (CBD) or opioids (including prescribed)
* Serious alcohol withdrawal symptoms as indicated by a score ≥ 10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised
* If female: pregnancy, nursing, or refusal to use reliable method of birth control; if using hormonal contraceptives, refusal to use secondary birth control method
* Any autoimmune or inflammatory medical disorder or medical condition that may interfere with safe study participation and/or study aims (e.g., unstable cardiac, renal, or liver disease, uncontrolled hypertension or diabetes)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or γ-glutamyl transferase (GGT) ≥ 4 times upper normal limit
* Attempted suicide in the past 3 years and/or serious suicidal intention or plan within the past year
* Currently on prescription medication that contraindicates use of minocycline, including but not necessarily limited to: isoretinoin, ergot alkaloids, and anti-coagulants.
* Previously known hypersensitivity to tetracyclines
* Current or recent (within one month) treatment with any antibiotic
* Regular use of a prebiotic or probiotic supplement
* Claustrophobia or physical issues preventing MRI scan
* Presence of a metal device in the body (e.g., pacemaker, infusion pump, aneurysm clip, metal prosthesis or plate)
* Current or recent (within 3 months) participation in a clinical trial involving medication administration
* Suffered a mild or moderate traumatic brain injury (TBI) within the last 12 months, a severe TBI at any point in their life, or a moderate TBI before the age of 12.
* Having below a 6th grade reading level
* Within the last 3 months, tested positive for COVID-19 (i.e. the SARS-CoV-2 virus) and experienced common related symptoms.
* Any other circumstances that, in the opinion of the investigators, compromises participant safety, ability of the investigators to conduct the study as designed, and/or study integrity.

Healthy Control Group Inclusion Criteria:

* Does not meet DSM-5 diagnostic criteria for an AUD (current or lifetime)
* In the 30-day period before enrollment, consume ≤ 14 and ≤ 7 standard drinks per week for men and women, respectively
* Engage in infrequent heavy drinking during the past 6 months (≤ 2 heavy drinking events in past 6 months)

Healthy Control Group Exclusion Criteria:

* Lifetime DSM-5 diagnosis of substance use disorder for any psychoactive substances other than nicotine
* Self-reported daily use of cannabidiol (CBD) or opioids (including prescribed)
* Lifetime DSM-5 diagnosis of schizophrenia spectrum and other psychotic disorders, bipolar and related disorders, depressive disorders, anxiety disorders (panic disorder, agoraphobia, social anxiety, and generalized anxiety), obsessive-compulsive and related disorders, trauma- and stressor-related disorders, feeding and eating disorders (binge eating, anorexia, and bulimia), conduct disorders, and gambling disorder
* Positive urine toxicology screen for the following substances: cocaine, opiates, amphetamines, methamphetamine, phencyclidine, barbiturates, benzodiazepine, methadone, and tricyclic antidepressants.
* Serious alcohol withdrawal symptoms as indicated by a score ≥ 10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised
* If female: pregnancy, nursing, or refusal to use reliable method of birth control; if using hormonal contraceptives, refusal to use secondary birth control method
* Any autoimmune or inflammatory medical disorder or medical condition that may interfere with safe study participation and/or study aims (e.g., unstable cardiac, renal, or liver disease, uncontrolled hypertension or diabetes)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or γ-glutamyl transferase (GGT) ≥ 4 times upper normal limit
* Attempted suicide in the past 3 years and/or serious suicidal intention or plan within the past year
* Currently on prescription medication that contraindicates use of minocycline, including but not necessarily limited to: isoretinoin, ergot alkaloids, and anti-coagulants.
* Previously known hypersensitivity to tetracyclines
* Current or recent (within one month) treatment with any antibiotic
* Regular use of a prebiotic or probiotic supplement
* Claustrophobia or physical issues preventing MRI scan
* Presence of a metal device in the body (e.g., pacemaker, infusion pump, aneurysm clip, metal prosthesis or plate)
* Current or recent (within 3 months) participation in a clinical trial involving medication administration
* Suffered a mild or moderate traumatic brain injury (TBI) within the last 12 months, a severe TBI at any point in their life, or a moderate TBI before the age of 12.
* Having below a 6th grade reading level
* Within the last 3 months, tested positive for COVID-19 (i.e. the SARS-CoV-2 virus) and experienced common related symptoms.
* Any other circumstances that, in the opinion of the investigators, compromises participant safety, ability of the investigators to conduct the study as designed, and/or study integrity.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Neuroinflammation | Change from baseline after 28 days of medication dosing
  A multimodal MRI approach consisting of Diffusion Tensor Imaging (DTI) with free water imaging and Magnetic Resonance Spectroscopy (MRS) will be utilized to assess neuroinflammation
Cue-Induced Alcohol Craving | Change from baseline after 28 days of medication dosing
  Participants will listen to a 5-minute guided cue exposure script, during which they are exposed to both a neutral and their preferred alcoholic beverage. Prior to beginning the paradigm and after each cue exposure participants will rate their alcohol craving using the "Alcohol Urge Questionnaire (AUQ)" and cigarette craving using the "Brief Questionnaire on Smoking Urges (BQSU)." Both scales range from 1 to 7 with higher scores reflecting more craving.
Alcohol consumption | Change from baseline after 28 days of medication dosing
  Total drinks consumed assessed using the Timeline Follow Back
Verbal Fluency/Language | Change from baseline after 28 days of medication dosing
  Wechsler Abbreviated Scale of Intelligence (WASI)-Vocabulary, WASI-Similarities, Verbal Fluency (Animals), with higher scores indicating greater intellectual ability.
Speed of processing | Change from baseline after 28 days of medication dosing
  Brief Assessment of Cognition in Schizophrenia (BACS)-Symbol Coding [scored by number of correct numerals (range: 0 -110)]
Speed of processing | Change from baseline after 28 days of medication dosing
  Trail Making Test: Part A (scored by time to complete test with lower scores being better)
Speed of processing | Change from baseline after 28 days of medication dosing
  Grooved Pegboard (scored as a sum of the total time, total number of drops, and the total number of pegs correctly placed in the board with higher scores corresponding to worse performance)
Working Memory | Change from baseline after 28 days of medication dosing
  Wechsler Memory Scale (WMS)-Spatial Span (scored up to 32 correct series), Letter-Number Span (scored up to 30 correct series)
Attention | Change from baseline after 28 days of medication dosing
  Continuous Performance Test
Problem Solving/Executive Functioning | Change from baseline after 28 days of medication dosing
  Wisconsin Card Sorting Test-64
Inhibition/Impulsivity | Change from baseline after 28 days of medication dosing
  Stop-Signal Reaction Time
Verbal Learning | Change from baseline after 28 days of medication dosing
  Hopkins Verbal Learning Test
Visual Learning | Change from baseline after 28 days of medication dosing
  Brief Visuospatial Memory Test [scoring is as follows, 1) Total recall: The sum of all valid items generated across learning trials 1-3, 2) Delayed recall: The number of valid items generated after a delay (trial 4), 3) Percent retained: Delayed recall score divided by the higher of trial 2 or 3 × 100, and 4) Recognition Discrimination Index: True positive responses minus false positive responses.]

SECONDARY OUTCOMES:
Peripheral Proinflammatory Marker levels | At baseline (day zero) and after 7, 14, and 21 and 28 days of medication dosing
  Serum level of inflammatory molecules
Alcohol Use Disorder Severity | At baseline (day zero) and after 28 days of medication dosing
  Symptom count from the alcohol module for the Structured Clinical Interview for DSM-5
Gut microbiota | At baseline (day zero) and after 7, 14, and 21 and 28 days of medication dosing
  Gut microbiota from stool samples using the following parameters: 1) diversity and evenness (Shannon, Simpson index) and 2) similarity (phylogenetic UniFrac distance, Jensen-Shannon divergence)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roche, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Maryland Psychiatric Research Center (MPRC) Treatment Research Program (TRP), Catonsville, Maryland, United States

REFERENCES:
- [Derived] Wheeler PB, Mackey CD, Moskal D, Brady DJ, Foster KT, Marks RM, Dickerson DL, Kelly DL, Bennett ME, Roche DJO. Religiosity and the relationship between sexual trauma, alcohol use, and sleep quality: a moderated mediation model. Alcohol Alcohol. 2025 May 14;60(4):agaf030. doi: 10.1093/alcalc/agaf030. PMID 40483726